CLINICAL TRIAL: NCT06905223
Title: A Pilot Study on the Efficacy of a Synbiotic Formula (MQU10) in Improving Mood and Well-being in Adults With Mild to Moderate Depressive Symptoms
Brief Title: A Pilot Study of Synbiotics in Adults With Depressive Symptoms
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: GenieBiome Limited (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: AM01 (GB)
Record Dates: First submitted 2025-03-25; First posted 2025-04-01 (Actual); Last update posted 2025-06-08 (Actual); Status verified 2025-06

CONDITIONS: Depressive Symptoms Mild to Moderate in Severity
Keywords: Depressive symptoms; Synbiotics; Adult Mood
MeSH Terms: conditions — Depression

STUDY DESIGN:
Intervention Model Description: All subjects will receive one sachet of MQU10 for 6 weeks
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- MQU10 (Experimental): Subjects will take 1 sachet of synbiotics formula (MQU10) daily for 6 weeks
  Interventions: Dietary Supplement: MQU10

INTERVENTIONS:
Dietary Supplement: MQU10 — MQU10 consists of a blend of food-grade probiotic strains (20 billion CFU daily) and prebiotic compounds.

SUMMARY:
This study aims to explore the efficacy and safety of a synbiotic formula (MQU10) in improving mood and well-being in adults with mild to moderate depressive symptoms.

DETAILED DESCRIPTION:
Major depression disorder (MDD) affects up to 20% of the population. In Hong Kong, one in seven suffered from mental health disorders with depressive disorder being one of the most frequent diagnoses. Depression is characterized by persistently low mood and loss of interest, possibly resulting from multifactorial factors including brain chemical abnormalities, genetics, stress, trauma and medical conditions. Current treatments for depression mainly include medication that alters neurotransmission in the brain and cognitive behavioural therapy to change cognitive distortions and their associated behaviours. However, there are side effects associated with the use of antidepressant medications as well as perceived stigma in receiving antidepressants and the uptake and accessibility of psychotherapy is extremely low. Thus, alternative therapeutic options are therefore needed to manage depression and its associated symptoms.

Emerging evidence suggests the important role of gut microbiota and gut-brain axis in mood regulation. In particular, there is high comorbidity among individuals with depression and gastrointestinal conditions such as irritable bowel syndrome and inflammatory bowel disease. There is also evidence suggesting that gut microbiota could produce metabolites and compounds with neuroactive and immunomodulatory properties. Previous studies have also supported the association between the dysbiosis of gut microbiota and affective disorders. Clinical trials on the use of microbiome-based therapeutics showed some efficacy in improving depression and insomnia. Gut microbiota modulation could be a novel therapeutic strategy for improving mood problems.

This pilot, single-arm study aims to explore the efficacy and safety of a synbiotic formula (MQU10), which is composed of food-grade probiotic strains and prebiotic compounds, in improving mood and well-being in adults with mild to moderate depressive symptoms.

ELIGIBILITY:
Inclusion Criteria:

* Individuals aged 18 or above
* Patient Health Questionnaire-9 (PHQ-9) score between 5 to 14
* Literate and can complete the self-report questionnaires
* Able to understand the consent and sign the informed consent form

Exclusion Criteria:

* Current diagnosis of substance abuse or dependence;
* A current or past history of bipolar disorder, manic or hypomanic episodes, schizophrenia, personality disorder, posttraumatic stress disorder (PTSD), intellectual disability, neurodegenerative disorders (e. g, Parkinson's disease) or organic mental disorder
* Requiring immediate psychiatric care (e. g, imminently suicidal subjects) or have attempted suicide in the past 3 months
* Use of antipsychotics, antidepressants or sedatives, unless on a stable dose in the last 4 weeks
* History of severe organ failure, renal failure on dialysis, HIV infection
* Active malignancy within 5 years
* History of major surgery on the gastrointestinal tract, except cholecystectomy and appendectomy in the past 5 years
* Night shift work
* History of antibiotic use within 4 weeks
* History of allergy to probiotics or lactose leading to a severe allergic reaction
* Known pregnancy or lactating

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2025-04-03 (Actual); Primary Completion 2026-03-25 (Estimated); Study Completion 2027-09-26 (Estimated)

PRIMARY OUTCOMES:
Proportions of subjects with improvement in condition, assessed by the Clinical Global Impression - Global Improvement Scale (CGI-I) at 6 weeks | 6 weeks
  The improvement in condition will be assessed by the Clinical Global Impression - Global Improvement Scale (CGI-I) at 6 weeks. It is a 7-point Likert scale. The clinician investigator will rate the improvement as 1 = very much improved, 2 = much improved, 3 = minimally improved, 4 = no change, 5 = minimally worse, 6 = much worse, and 7 = very much worse.

SECONDARY OUTCOMES:
Self-report improvement in condition, assessed by Patient Global Impression of Change scale (PGI-C) by 6 weeks | 6 weeks
  The self-report improvement in condition will be assessed by Patient Global Impression of Change scale (PGI-C). It is a 7-point Likert scale. Subjects will rate their change as 1 = very much improved, 2 = much improved, 3 = minimally improved, 4 = no change, 5 = minimally worse, 6 = much worse, and 7 = very much worse.
Changes in depression level, assessed by Patient Health Questionnaire-9 (PHQ-9) by 6 weeks | 6 weeks
  Patient Health Questionnaire-9 (PHQ-9) is a 9-item instrument to assess the severity of depressive symptoms. Total score categories for PHQ-9 are 0-4 = minimal/no depression, 5-9 = mild depression, 10-14 = moderate depression, 15-19 = moderately severe depression, and 20-27 = severe depression.
Changes in anxiety level, assessed by Generalised Anxiety Disorder 7-item scale (GAD-7) by 6 weeks | 6 weeks
  Generalised Anxiety Disorder 7-item scale (GAD-7) consists of seven questions that measure the frequency and intensity of anxiety symptoms experienced over the past two weeks. The total score on the GAD-7 can range from 0 to 21, with higher scores indicating more severe anxiety symptoms
Changes in health-related quality of life, assessed by World Health Organization Quality of Life-BREF (WHOQOL-BREF) by 6 weeks | 6 weeks
  World Health Organization Quality of Life-BREF (WHOQOL-BREF) is a 26-item self-report instrument consisting of four domains: physical health, psychological health, social relationships, and environmental health, with quality of life and general health items. Each item is scored on a five-point scale, and the scores are transformed linearly to a 0-100 scale
Changes in gut microbiota composition and functions by 6 weeks | 6 weeks
  The changes of microbial profile in stool compared to baseline
Adverse events by 6 weeks | 6 weeks
  The adverse events reported throughout the study

CONTACTS AND LOCATIONS:
Overall Officials: Jessica Ching, PhD, Study Director — GenieBiome Limited
Locations (2):
- Hong Kong (2):
  - GenieBiome Limited, Hong Kong
  - Healthymind Centre, Hong Kong

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Yong SJ, Tong T, Chew J, Lim WL. Antidepressive Mechanisms of Probiotics and Their Therapeutic Potential. Front Neurosci. 2020 Jan 14;13:1361. doi: 10.3389/fnins.2019.01361. eCollection 2019. PMID 32009871
- [Background] Poluektova E, Yunes R, Danilenko V. The Putative Antidepressant Mechanisms of Probiotic Bacteria: Relevant Genes and Proteins. Nutrients. 2021 May 10;13(5):1591. doi: 10.3390/nu13051591. PMID 34068669
- [Background] Huang R, Wang K, Hu J. Effect of Probiotics on Depression: A Systematic Review and Meta-Analysis of Randomized Controlled Trials. Nutrients. 2016 Aug 6;8(8):483. doi: 10.3390/nu8080483. PMID 27509521
- [Background] Lau RI, Su Q, Lau ISF, Ching JYL, Wong MCS, Lau LHS, Tun HM, Mok CKP, Chau SWH, Tse YK, Cheung CP, Li MKT, Yeung GTY, Cheong PK, Chan FKL, Ng SC. A synbiotic preparation (SIM01) for post-acute COVID-19 syndrome in Hong Kong (RECOVERY): a randomised, double-blind, placebo-controlled trial. Lancet Infect Dis. 2024 Mar;24(3):256-265. doi: 10.1016/S1473-3099(23)00685-0. Epub 2023 Dec 7. PMID 38071990
- [Background] Pirbaglou M, Katz J, de Souza RJ, Stearns JC, Motamed M, Ritvo P. Probiotic supplementation can positively affect anxiety and depressive symptoms: a systematic review of randomized controlled trials. Nutr Res. 2016 Sep;36(9):889-898. doi: 10.1016/j.nutres.2016.06.009. Epub 2016 Jun 21. PMID 27632908
- [Background] Ito H, Tomura Y, Kitagawa Y, Nakashima T, Kobanawa S, Uki K, Oshida J, Kodama T, Fukui S, Kobayashi D. Effects of probiotics on sleep parameters: A systematic review and meta-analysis. Clin Nutr ESPEN. 2024 Oct;63:623-630. doi: 10.1016/j.clnesp.2024.07.006. Epub 2024 Aug 2. PMID 39094854
- [Background] Gil-Hernandez E, Ruiz-Gonzalez C, Rodriguez-Arrastia M, Ropero-Padilla C, Rueda-Ruzafa L, Sanchez-Labraca N, Roman P. Effect of gut microbiota modulation on sleep: a systematic review and meta-analysis of clinical trials. Nutr Rev. 2023 Nov 10;81(12):1556-1570. doi: 10.1093/nutrit/nuad027. PMID 37023468
- [Background] Li Y, Hao Y, Fan F, Zhang B. The Role of Microbiome in Insomnia, Circadian Disturbance and Depression. Front Psychiatry. 2018 Dec 5;9:669. doi: 10.3389/fpsyt.2018.00669. eCollection 2018. PMID 30568608
- [Background] Matenchuk BA, Mandhane PJ, Kozyrskyj AL. Sleep, circadian rhythm, and gut microbiota. Sleep Med Rev. 2020 Oct;53:101340. doi: 10.1016/j.smrv.2020.101340. Epub 2020 May 13. PMID 32668369
- [Background] Haarhuis JE, Kardinaal A, Kortman GAM. Probiotics, prebiotics and postbiotics for better sleep quality: a narrative review. Benef Microbes. 2022 Aug 3;13(3):169-182. doi: 10.3920/BM2021.0122. Epub 2022 Jul 11. PMID 35815493
- [Background] Cryan JF, Dinan TG. Mind-altering microorganisms: the impact of the gut microbiota on brain and behaviour. Nat Rev Neurosci. 2012 Oct;13(10):701-12. doi: 10.1038/nrn3346. Epub 2012 Sep 12. PMID 22968153
- [Background] Clapp M, Aurora N, Herrera L, Bhatia M, Wilen E, Wakefield S. Gut microbiota's effect on mental health: The gut-brain axis. Clin Pract. 2017 Sep 15;7(4):987. doi: 10.4081/cp.2017.987. eCollection 2017 Sep 15. No abstract available. PMID 29071061
- [Background] Brown JSL. Increasing access to psychological treatments for adults by improving uptake and equity: rationale and lessons from the UK. Int J Ment Health Syst. 2018 Nov 9;12:67. doi: 10.1186/s13033-018-0246-7. eCollection 2018. PMID 30455729
- [Background] Bet PM, Hugtenburg JG, Penninx BW, Hoogendijk WJ. Side effects of antidepressants during long-term use in a naturalistic setting. Eur Neuropsychopharmacol. 2013 Nov;23(11):1443-51. doi: 10.1016/j.euroneuro.2013.05.001. Epub 2013 May 30. PMID 23726508
- [Background] Lam LC, Wong CS, Wang MJ, Chan WC, Chen EY, Ng RM, Hung SF, Cheung EF, Sham PC, Chiu HF, Lam M, Chang WC, Lee EH, Chiang TP, Lau JT, van Os J, Lewis G, Bebbington P. Prevalence, psychosocial correlates and service utilization of depressive and anxiety disorders in Hong Kong: the Hong Kong Mental Morbidity Survey (HKMMS). Soc Psychiatry Psychiatr Epidemiol. 2015 Sep;50(9):1379-88. doi: 10.1007/s00127-015-1014-5. Epub 2015 Feb 8. PMID 25660760
- [Background] Kessler RC, Chiu WT, Demler O, Merikangas KR, Walters EE. Prevalence, severity, and comorbidity of 12-month DSM-IV disorders in the National Comorbidity Survey Replication. Arch Gen Psychiatry. 2005 Jun;62(6):617-27. doi: 10.1001/archpsyc.62.6.617. PMID 15939839